CLINICAL TRIAL: NCT06111612
Title: Intensive Conditioning Regimen With Thiotepa Combined With Busulfan, Fludarabine and Cytarabine for Allogeneic Hematopoietic Stem Cell Transplantation in the Treatment of Myeloid Malignancies With Extramedullary Involvement
Brief Title: Intensive Conditioning withTHI/Bu/Flu/Ara-C in Allo-HSCT for Myeloid Malignancies With Extramedullary Involvement
Status: Recruiting | Type: Observational
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Xianmin Song, MD, Professor, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Other Study IDs: SHSYXY-202308-THI-BFA
Record Dates: First submitted 2023-10-27; First posted 2023-11-01 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Neoplasm; Chronic Myelomonocytic Leukemia; Myeloid Sarcoma; Extramedullary Myeloid Tumor
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Anemia, Refractory, with Excess of Blasts; Leukemia, Myelomonocytic, Chronic; Sarcoma, Myeloid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
This study is a multicenter, single-arm, prospective phase II clinical trial that evaluates the efficacy and safety of an intensive conditioning regimen with thiotepa combined with busulfan, fludarabine, and cytarabine for allogeneic hematopoietic stem cell transplantation in the treatment of myeloid malignancies with extramedullary involvement. The conditioning regimen includes thiotepa at a dose of 5mg/kg/d from d -9 to d -8 (2 days), fludarabine at 30mg/m2/d from d -7 to d -3 (5 days), cytarabine at 1-1.5g/m2/d from d -7 to d -3 (5 days), and busulfan at 3.2mg/kg/d from d -5 to d -3 (3 days). Conditioning begins on day -9, and donor hematopoietic stem cell infusion is performed on day 0. All patients will undergo bone marrow examination on day 14 and day 28 post-transplant, followed by bone marrow examinations every 30 days within the first year after transplantation, and every 60 days within the second year after transplantation. If disease relapse is suspected during the follow-up period, bone marrow or extramedullary relapse site examinations will be conducted at any time. The primary study endpoints are the 1-year and 2-year progression-free survival (PFS) rates post-transplant. Secondary study endpoints include the incidence of acute graft-versus-host disease (GVHD) within 180 days post-transplant, cumulative relapse rates at 1 year and 2 years post-transplant, 1-year and 2-year overall survival (OS), graft-versus-host disease-free, relapse-free survival (GRFS), non-relapse mortality (NRM), cumulative incidence of chronic GVHD, and the incidence of Cytomegalovirus （CMV）and Epstein-Barr virus（EBV）reactivation within 1 year.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and less than 55 years, regardless of gender.
2. Criteria for myeloid tumors with extramedullary involvement:

   1. AML (Acute Myeloid Leukemia) with at least one extramedullary lesion achieving hematological remission (CR1 or CR2) after induction therapy.
   2. MDS (Myelodysplastic Syndrome) with at least one extramedullary lesion and bone marrow blast percentage ≥ 5% achieving hematological CR after treatment; CMML (Chronic Myelomonocytic Leukemia) with at least one extramedullary lesion (diagnosed according to WHO standards) achieving hematological CR after treatment.
   3. Control and remission of extramedullary lesions, including those in the central nervous system, testes, skin, and other extramedullary tissues.
   4. Granulocytic sarcoma with or without bone marrow involvement, and achieving remission after treatment.
3. Patients must have a suitable hematopoietic stem cell donor:

   1. Related donors must have at least 5/10 matches for HLA-A, -B, -C, -DQB1, and - DRB1.
   2. Unrelated donors must have at least 8/10 matches for HLA-A, -B, -C, -DQB1, and

      * DRB1.
4. Hematopoietic cell transplantation comorbidity index (HCT-CI) score ≤ 2.
5. ECOG (Eastern Cooperative Oncology Group) performance status: 0-2.
6. Adequate liver, kidney, and cardiopulmonary function, meeting the following requirements:

   1. Serum creatinine ≤ 1.5x ULN (the upper limit of normal).
   2. Cardiac function: Ejection fraction ≥ 50%.
   3. Baseline oxygen saturation > 92%.
   4. Total bilirubin ≤ 1.5 x ULN; ALT and AST ≤ 2.0 x ULN.
   5. Pulmonary function: DLCO (corrected for hemoglobin) ≥ 40% and FEV1 (Forced Expiratory Volume in 1 second) ≥ 50%.
7. Patients must have the ability to understand and be willing to participate in this study and sign an informed consent form.

Exclusion Criteria:

1. History of malignancies other than myeloid tumors within the 5 years prior to screening, except for adequately treated in situ cervical cancer, basal cell carcinoma, squamous cell carcinoma of the skin, and curatively treated localized prostate cancer or ductal carcinoma in situ.
2. ECOG > 2.
3. HCT-CI score ≥ 3.
4. Any unstable systemic diseases, including but not limited to unstable angina, recent cerebrovascular accidents or transient ischemic attacks within the 3 months prior to screening, myocardial infarction within the 3 months prior to screening, congestive heart failure (New York Heart Association [NYHA] class ≥ III), severe arrhythmias requiring drug treatment after pacemaker implantation, significant liver, kidney, or metabolic diseases, and pulmonary arterial hypertension.
5. Active, uncontrolled infections, including those associated with hemodynamic instability, new or worsening infection symptoms or signs, new infectious lesions on imaging, or persistent unexplained fever without signs or symptoms of infection.
6. Conditions requiring treatment such as grade 2 or higher seizures, paralysis, aphasia, recent severe cerebral infarction, severe traumatic brain injury, dementia, Parkinson's disease, or schizophrenia.
7. HIV-infected individuals.
8. Active hepatitis B (HBV) or active hepatitis C (HCV) requiring antiviral therapy.

   Patients at risk of HBV reactivation, are defined as those who are positive for hepatitis B surface antigen or core antibody without receiving antiviral therapy.
9. Pregnant or breastfeeding women.
10. Fertile males and females unwilling to use contraception during the treatment period and for 12 months after treatment.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Outpatient and inpatient patients
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-01-20 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
1y and 2y-PFS | 2023-2027
  1-year and 2-year progression-free survival (PFS) rates post-transplant

SECONDARY OUTCOMES:
aGVHD | 2023-2025
  acute graft-versus-host disease (GVHD) within 180 days post-transplant
1y and 2y-CIR | 2023-2027
  cumulative relapse rates (CIR) at 1 year and 2 years post-transplant
1y and 2y-OS | 2023-2027
  overall survival (OS) at 1 year and 2 years post-transplant
GRFS | 2023-2027
  graft-versus-host disease-free, relapse-free survival (GRFS) at 2 years post-transplant
NRM | 2023-2027
  non-relapse mortality (NRM) at 2 years post-transplant
cGVHD | 2023-2027
  cumulative incidence of chronic GVHD at 2 years post-transplant
CMV and EBV reactivation | 2023-2026
  the incidence of CMV and EBV reactivation within 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Xianmin Song, MD, Principal Investigator — Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Shanghai General Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Martin-Subero JI. Predicting leukemia relapse. Nat Med. 2018 Apr 10;24(4):385-387. doi: 10.1038/nm.4529. No abstract available. PMID 29634681
- [Background] Elenitoba-Johnson K, Hodges GF, King TC, Wu CD, Medeiros LJ. Extramedullary myeloid cell tumors arising in the setting of chronic myelomonocytic leukemia. A report of two cases. Arch Pathol Lab Med. 1996 Jan;120(1):62-7. PMID 8554447
- [Background] Hancock JC, Prchal JT, Bennett JM, Listinsky CM. Trilineage extramedullary myeloid cell tumor in myelodysplastic syndrome. Arch Pathol Lab Med. 1997 May;121(5):520-3. PMID 9167610
- [Background] Cankaya H, Ugras S, Dilek I. Head and neck granulocytic sarcoma with acute myeloid leukemia: three rare cases. Ear Nose Throat J. 2001 Apr;80(4):224-6, 228-9. PMID 11338646
- [Background] Bakst RL, Tallman MS, Douer D, Yahalom J. How I treat extramedullary acute myeloid leukemia. Blood. 2011 Oct 6;118(14):3785-93. doi: 10.1182/blood-2011-04-347229. Epub 2011 Jul 27. PMID 21795742
- [Background] Cribe AS, Steenhof M, Marcher CW, Petersen H, Frederiksen H, Friis LS. Extramedullary disease in patients with acute myeloid leukemia assessed by 18F-FDG PET. Eur J Haematol. 2013 Apr;90(4):273-8. doi: 10.1111/ejh.12085. PMID 23470093
- [Background] Su WP. Clinical, histopathologic, and immunohistochemical correlations in leukemia cutis. Semin Dermatol. 1994 Sep;13(3):223-30. PMID 7986692
- [Background] Pileri SA, Ascani S, Cox MC, Campidelli C, Bacci F, Piccioli M, Piccaluga PP, Agostinelli C, Asioli S, Novero D, Bisceglia M, Ponzoni M, Gentile A, Rinaldi P, Franco V, Vincelli D, Pileri A Jr, Gasbarra R, Falini B, Zinzani PL, Baccarani M. Myeloid sarcoma: clinico-pathologic, phenotypic and cytogenetic analysis of 92 adult patients. Leukemia. 2007 Feb;21(2):340-50. doi: 10.1038/sj.leu.2404491. Epub 2006 Dec 14. PMID 17170724
- [Background] Chevallier P, Mohty M, Lioure B, Michel G, Contentin N, Deconinck E, Bordigoni P, Vernant JP, Hunault M, Vigouroux S, Blaise D, Tabrizi R, Buzyn A, Socie G, Michallet M, Volteau C, Harousseau JL. Allogeneic hematopoietic stem-cell transplantation for myeloid sarcoma: a retrospective study from the SFGM-TC. J Clin Oncol. 2008 Oct 20;26(30):4940-3. doi: 10.1200/JCO.2007.15.6315. Epub 2008 Jul 7. PMID 18606981
- [Background] Michel G, Boulad F, Small TN, Black P, Heller G, Castro-Malaspina H, Childs BH, Gillio AP, Papadopoulos EB, Young JW, Kernan NA, O'Reilly RJ. Risk of extramedullary relapse following allogeneic bone marrow transplantation for acute myelogenous leukemia with leukemia cutis. Bone Marrow Transplant. 1997 Jul;20(2):107-12. doi: 10.1038/sj.bmt.1700857. PMID 9244412
- [Background] Pui CH, Kalwinsky DK, Schell MJ, Mason CA, Mirro J Jr, Dahl GV. Acute nonlymphoblastic leukemia in infants: clinical presentation and outcome. J Clin Oncol. 1988 Jun;6(6):1008-13. doi: 10.1200/JCO.1988.6.6.1008. PMID 3373258
- [Background] Bruserud O, Reikvam H, Kittang AO, Ahmed AB, Tvedt TH, Sjo M, Hatfield KJ. High-dose etoposide in allogeneic stem cell transplantation. Cancer Chemother Pharmacol. 2012 Dec;70(6):765-82. doi: 10.1007/s00280-012-1990-z. Epub 2012 Oct 6. PMID 23053272
- [Background] Clift RA, Buckner CD, Appelbaum FR, Sullivan KM, Storb R, Thomas ED. Long-term follow-Up of a randomized trial of two irradiation regimens for patients receiving allogeneic marrow transplants during first remission of acute myeloid leukemia. Blood. 1998 Aug 15;92(4):1455-6. No abstract available. PMID 9694737
- [Background] Alatrash G, de Lima M, Hamerschlak N, Pelosini M, Wang X, Xiao L, Kerbauy F, Chiattone A, Rondon G, Qazilbash MH, Giralt SA, de Padua Silva L, Hosing C, Kebriaei P, Zhang W, Nieto Y, Saliba RM, Champlin RE, Andersson BS. Myeloablative reduced-toxicity i.v. busulfan-fludarabine and allogeneic hematopoietic stem cell transplant for patients with acute myeloid leukemia or myelodysplastic syndrome in the sixth through eighth decades of life. Biol Blood Marrow Transplant. 2011 Oct;17(10):1490-6. doi: 10.1016/j.bbmt.2011.02.007. Epub 2011 Feb 18. PMID 21338705
- [Background] Sora F, Grazia CD, Chiusolo P, Raiola AM, Bregante S, Mordini N, Olivieri A, Iori AP, Patriarca F, Grisariu S, Terruzzi E, Rambaldi A, Sica S, Bruno B, Angelucci E, Bacigalupo A. Allogeneic Hemopoietic Stem Cell Transplants in Patients with Acute Myeloid Leukemia (AML) Prepared with Busulfan and Fludarabine (BUFLU) or Thiotepa, Busulfan, and Fludarabine (TBF): A Retrospective Study. Biol Blood Marrow Transplant. 2020 Apr;26(4):698-703. doi: 10.1016/j.bbmt.2019.12.725. Epub 2019 Dec 23. PMID 31875522
- [Background] Down JD, Westerhof GR, Boudewijn A, Setroikromo R, Ploemacher RE. Thiotepa improves allogeneic bone marrow engraftment without enhancing stem cell depletion in irradiated mice. Bone Marrow Transplant. 1998 Feb;21(4):327-30. doi: 10.1038/sj.bmt.1701103. PMID 9509964
- [Background] Li C, Mathews V, Kim S, George B, Hebert K, Jiang H, Li C, Zhu Y, Keesler DA, Boelens JJ, Dvorak CC, Agarwal R, Auletta JJ, Goyal RK, Hanna R, Kasow K, Shenoy S, Smith AR, Walters MC, Eapen M. Related and unrelated donor transplantation for beta-thalassemia major: results of an international survey. Blood Adv. 2019 Sep 10;3(17):2562-2570. doi: 10.1182/bloodadvances.2019000291. PMID 31471325
- [Background] Sanders S, Chua N, Larouche JF, Owen C, Shafey M, Stewart DA. Outcomes of Consecutively Diagnosed Primary Central Nervous System Lymphoma Patients Using the Alberta Lymphoma Clinical Practice Guideline Incorporating Thiotepa-Busulfan Conditioning for Transplantation-Eligible Patients. Biol Blood Marrow Transplant. 2019 Aug;25(8):1505-1510. doi: 10.1016/j.bbmt.2019.04.004. Epub 2019 Apr 6. PMID 30965138